CLINICAL TRIAL: NCT04049526
Title: The Effects of Different Music Genres on Heart Rate Variability in Extremely and Very Low Birth Weight Premature Newborns: An Italian Pilot Study
Brief Title: The Effects of Different Music Genres on Heart Rate Variability in Extremely and Very Low Birth Weight Newborns
Status: Completed | Type: Observational
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Barbara Sgobbi, Musicotherapist, Ospedale di Circolo - Fondazione Macchi
Other Study IDs: 51
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Infant Behavior; Infant Conditions; Infant Morbidity
Keywords: Music; Preterm infants; Heart Rate Variability
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: The influence of different music genres on Heart Rate Variability (HRV) in preterm infants — Neonates undergo a daily randomized music listening program (25 minutes, every day, for 3 days) based on different music genres listening (soft pop-rap, pop-rock and classical music). Music programs is followed by 1 day of no music monitoring (25 minutes). An electrocardiogram is performed to evaluate HRV parameters in each neonate with and without music exposure

SUMMARY:
AIM: to investigate the influence of different music genres on Heart Rate Variability (HRV) of preterm infants.

Neonates undergo a daily randomized music listening program. An electrocardiogram is performed to evaluate HRV parameters in each neonate with and without music exposure.

DETAILED DESCRIPTION:
AIM: to investigate the influence of different music genres on Heart Rate Variability (HRV) of preterm infants.

HRV has been previously used to evaluate autonomic nervous system fluctuations in heart rate related to maturation in healthy neonates and in neonates with pathological conditions. This parameter has been used to show how music could improve well-being and the development of the autonomic nervous system in infants.

In this study, neonates (see also inclusion/exclusion criteria), recruited on the basis of birth order, undergo a daily randomized music listening program (25 minutes, every day, for 3 days) based on different music genres listening (soft pop-rap, pop-rock and classical music). Music programs is followed by 1 day of no music monitoring (25 minutes). An electrocardiogram is performed to evaluate HRV parameters in each neonate with and without music exposure.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between the 23th and the 32nd week
* birth weight <1500g
* appropriate for gestational age, sufficient stability of the vital parameters and absence of active infections and episodes of apnoea during the 72 hours before the test

Exclusion Criteria:

* genetic anomalies, chromosomal aberrations, congenital heart malformations, intraventricular haemorrhage (> grade II on ultrasound), periventricular Leukomalacia
* neonates with failed responses to bilateral hearing screening performed by Automated Auditory Brainstem Response testing

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Enrollment performed when sufficient stability of the vital parameters and absence of active infections and episodes of apnoea during the 72 hours before the test
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) variation in preterm infants according to different music genres listening | Enrollment performed when sufficient stability of the vital parameters and absence of active infections and episodes of apnoea during the 72 hours before the treatment
  An electrocardiogram is performed to evaluate HRV parameters in each neonate with and without music exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sgobbi, Principal Investigator — Tincontro Onlus
Locations (1):
- Barbara Sgobbi, Varese, Italy